CLINICAL TRIAL: NCT05504538
Title: The Correlation Between Coracoid Tunnel Dilatation and Loss of Reduction After Arthroscopic Acromioclavicular Fixation Using Tightrope System, A CT Based Study
Brief Title: Coracoid Tunnel Widening After ACJ Tight Rope Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Refaat Waly, Principal investigator, Consultant of Trauma and Orthopedics, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-170518
Record Dates: First submitted 2022-08-02; First posted 2022-08-17 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Orthopedic Disorder; Orthopedic Devices Associated With Misadventures
Keywords: Acute acromioclavicular joint injury .; TightRope .; Coracoid tunnel dilatation.; Loss of reduction.
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- patient with Acute acromioclavicular joint injury (Experimental): patient with Acute acromioclavicular joint injury
  Interventions: Procedure: arthroscopic fixation of Acute acromioclavicular joint injury using tight rope; Device: Tight rope

INTERVENTIONS:
Procedure: arthroscopic fixation of Acute acromioclavicular joint injury using tight rope — arthroscopic fixation of Acute acromioclavicular joint injury using tight rope
Device: Tight rope — Adjustable button device from Arthrex Naples USA

SUMMARY:
studying coracoid tunnel widening after arthroscopic fixation of acute acromioclavicular joint (ACJ) dislocation using TightRope system and its correlation with loss of reduction and the functional scores.

DETAILED DESCRIPTION:
Abstract Purpose: To detect coracoid tunnel widening after arthroscopic fixation of acute acromioclavicular joint (ACJ) dislocation using TightRope system and its correlation with loss of reduction and the functional scores.

Methods: From July 2016 to Dec 2018, a prospective study was performed at our hospital. Twenty-three patients with acute grade III-V ACJ dislocation were included in the study. Arthroscopic double tight-rope repair of the ACJ was performed. Coracoid tunnel widening was measured by computed tomography (CT) and coraco-clavicular distance was measured on the x-ray immediately post-operative and at 12 months. Constant Shoulder Score, Oxford Shoulder Score, Nottingham Clavicle Score and Visual analogue scale were used as outcome measures at 12 months.

Level of evidence IV Keywords Acute acromioclavicular joint injury . TightRope . Coracoid tunnel dilatation. Loss of reduction.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute (≤ 3 weeks after injury) Rockwood grade III-V ACJ dislocation

Exclusion Criteria:

* Patients with associated coracoid fracture, associated rotator cuff tears or glenohumeral arthritis

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Coracoid tunnel diameter difference between immediate postoperative and final follow up | 1 year
  Radiological outcome using CT scans
Coraco-clavicular distance immediate postoperative and at final follow up | 1 year
  Radiological outcome using X-rays

SECONDARY OUTCOMES:
Constant-Murley shoulder score. Ranges from 0 representing worst outcome to 100 representing best outcome | 1 year
  Clinical score using a questionnaire
Disability of arm shoulder and Hand score ( DASH score) highest is 100 which represents worst outcome while lowest is 0 representing best possible outcome | 1 year
  Clinical score using a questionnaire
Oxford Shoulder score, a questionnaire of 12 questions each scores from 1 to 5. 1 being the fewest symptoms, 5 being the worst. The total score is 60 marks, the higher the score the worse the outcomes | 1 year
  Clinical score using a questionnaire

IPD SHARING:
Plan to Share IPD: No